CLINICAL TRIAL: NCT06079437
Title: The Effect of Brief Skin Cooling on Isometric Muscle Strength and the Neuronal Mechanism Underlying This Effect
Brief Title: The Effect of Brief Skin Cooling on Isometric Muscle Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mert Cetin, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CISVWSA
Record Dates: First submitted 2023-09-29; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Cryotherapy Effect
Keywords: soleus v-wave; sympathetic outflow; muscle spindle; cold stress test; sympathetic system; contractile force; motor facilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Heart rate, maximum isometric muscle strength, Soleus H-reflex, M-wave, and V-wave measurements were taken in three consecutive periods. First-period maximal isometric contraction; second-period maximal isometric contraction + cold pressure test; third-period maximal isometric contraction + Cheering
  Interventions: Procedure: Cheer; Procedure: The cold pressure test

INTERVENTIONS:
Procedure: Cheer — Maximum isometric contraction was performed with cheering.
Procedure: The cold pressure test — Maximum isometric contraction was performed with the cold pressure test.

SUMMARY:
There is sympathetic innervation of the muscular spindle. The application of cold to the skin provides an increase in sympathetic activity. In rehabilitation practice, short-term local cold is applied to the skin to provide motor facilitation. The aim of this study was to examine whether short-term local cold application provides an increase in isometric contractile strength and, if so, whether this effect is related to muscle spindle activity.

DETAILED DESCRIPTION:
Cold application is frequently used in sports medicine and rehabilitation due to its beneficial effects on the neuromuscular system. Its main beneficial effects are facilitating muscle contraction (motor facilitation), increasing isometric muscle force formation and reducing spasticity. The motor effects of cold application may vary depending on the application time, cooling agent (ice, ice water, cooling spray, etc.) and subcutaneous fatty tissue thickness. Short-term cold application can increase contraction force through motor facilitation. As the duration of cold application increases, the effects of cold that inhibit motor functions, such as gamma motor neuron inhibition, muscle spindle inhibition, and muscle conduction block, come to the fore. With this effect, it is used in the treatment of spasticity.

Neurophysiological studies to explain the motor effects of cold application have generally focused on the monosynaptic muscle spindle-based reflex. The monosynaptic muscle spindle-based reflex activates muscle spindles and stimulates alpha motor neurons via Group Ia afferent nerves. This effect is also known as the servo-motor (servo-assistance) effect of the muscle spindle. The increase in the sensitivity of the muscle spindle can provide motor facilitation by strengthening the servo-assistance effect.

It has been shown that the muscle spindle has sympathetic innervation. It has been shown that the cold stress test can be an alternative to the classical autonomic nerve test and can be used to test sympathetic system activation. Additionally, studies have shown that cold stress test, mental arithmetic, isometric contraction and muscle ischemia cause an increase in muscle spindle sensitivity through increased sympathetic activity.

A literature review has shown that there is no study examining the mechanism underlying the effect of local cold application on motor facilitation. Demonstrating the effect of local cold application on increasing maximum contraction force through muscle spindle sensitivity is also important for clinical applications to be more effective and efficient. The aim of this study was to examine whether short-term local cold application increases isometric contraction force and, if there is an increase, whether this effect is related to muscle spindle activity.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy
* Being a young adult (20-45 years old)
* Volunteer

Exclusion Criteria:

* Scar, dermatitis, etc. in the skin tissue where the surface electromyography electrode will be placed
* Upper extremity bone and joint disease, history of neuromuscular disease
* Heart disease, Hypertension
* Cold intolerance

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-22 (Actual)

PRIMARY OUTCOMES:
Heart rate | during procedure
  Heart rate was monitored with DII derivation electrocardiographic recording. Heart rate was reported as beats per minute.
Soleus H-reflex amplitude | during procedure
  By stimulating the tibial nerve with an electrical current, the Soleus H-reflex was obtained. Its peak to peak amplitude will be measured in microvolts.
Soleus V-wave amplitude | during procedure
  Soleus V-wave was obtained by applying an electrical current to the tibial nerve during maximum voluntary contraction (MCV). Peak-to-peak amplitude was measured in microvolts.
Maximum isometric muscle strength | during procedure
  Maximum isometric muscle strength of ankle plantar flexors was measured using a force sensor

SECONDARY OUTCOMES:
Skin temperature | during procedure
  The skin temperature of the back of the hand exposed to the cold application was measured with an infrared thermometer and the results were reported in degrees Celsius.

CONTACTS AND LOCATIONS:
Overall Officials: Mert Cetin, MD, Principal Investigator — İstanbul Physical Therapy Rehabilitation Training & Research Hosptial
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training & Research Hospital, Istanbul, Turkey (Türkiye)